CLINICAL TRIAL: NCT02837965
Title: Multicenter Prospective Observational Study Assessing Outcomes, Adverse Events, Treatment Patterns and Related Costs in Patients Diagnosed With Bullous Pemphigoid
Brief Title: Observational Study Assessing Outcomes, Treatment Patterns and Related Costs in Patients in Bullous Pemphigoid
Acronym: EDP-PB
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PR12042*
Record Dates: First submitted 2016-06-24; First posted 2016-07-20 (Estimated); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Bullous Pemphigoid
MeSH Terms: conditions — Pemphigoid, Bullous | interventions — Therapeutics; Methotrexate; Prednisone; Doxycycline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- diagnosed bullous pemphigoid
  Interventions: Drug: treatment with topical superpotent corticosteroid therapy; Drug: treatment with systemic therapy (methotrexate); Drug: treatment systemic therapy (prednisone); Drug: treatment with systemic therapy (prednisone); Drug: treatment with systemic therapy (doxycycline)

INTERVENTIONS:
Drug: treatment with topical superpotent corticosteroid therapy
Drug: treatment with systemic therapy (methotrexate)
Drug: treatment systemic therapy (prednisone)
Drug: treatment with systemic therapy (prednisone)
Drug: treatment with systemic therapy (doxycycline)

SUMMARY:
The study is an observational, multi-center, prospective, non-interventional and open-label data collection study assessing outcomes, treatment patterns, adverse events and costs in patients diagnosed with bullous pemphigoid. The patient enrollment period will be 1 year with a follow-up (observation period) of 1 year for each patient. Four dermatology centres in France will participate. The hypothesis to be answered by the study is that superpotent topical corticosteroid therapy is properly used to treat bullous pemphigoid in real-world life as recommended by French guidelines and whether this treatment influences the medical costs by comparison with systemic therapies (e.g. methotrexate or prednisone).

DETAILED DESCRIPTION:
Bullous pemphigoid is the most common autoimmune blistering disease of the skin, usually affecting the elderly. It is a chronic disease characterized by spontaneous exacerbations and remissions. Bullous pemphigoid is mediated by IgG autoantibodies directed against hemidesmosomal proteins (BP180, BP230), which are involved in dermal-epidermal adhesion in the skin. The diagnosis of bullous pemphigoid is based on clinical and immunopathological findings, including skin direct immunofluorescence. The disease usually requires on average a 1-year duration of treatment although a long-term maintenance therapy may be necessary some cases. High doses oral corticosteroids have been considered as the mainstay of treatment for many years, but are deleterious, with a high rate of treatment side effects, including mortality. Topical superpotent corticosteroids have been demonstrated to be as effective but safer than high doses of oral corticosteroids, reducing side effects and mortality rate, while controlling the disease in between 95% to 100% of cases. Despite its high efficacy, topical superpotent corticosteroid therapy is often considered as poorly convenient. In addition, immunosuppressant drugs and methotrexate are poorly tolerated or frequently contra-indicated in those elderly patients with bullous pemphigoid. To date, no study has evaluated the real-world use and costs of the different treatments in this disease.

Purpose The project is an observational, multi-center, prospective, non-interventional and open-label data collection study assessing outcomes, adverse events, treatment patterns and related costs in patients diagnosed with bullous pemphigoid. The patient enrollment period will be 1 year with a follow-up (observation period) of 1 year for each patient. Four dermatology centres in France will participate.

Primary objective:

The specific goal is to describe in each patient with bullous pemphigoid the therapeutic management, including: i) all topical and systemic medications and nursing cares; ii) clinical and biological monitoring and iii) clinical outcome during the first year of treatment. The hypothesis to be answered by the study is that topical superpotent corticosteroid therapy is properly used to treat bullous pemphigoid in real-world life as recommended by French guidelines and whether this treatment influences the medical costs by comparison with systemic therapies (e.g. methotrexate or prednisone).

Secondary objectives:

* To determine the factors influencing the first-line therapy : topical superpotent corticosteroid therapy (treatment scheme 1 or TS1) versus systemic therapy (treatment scheme 2 or TS2).
* To determine the factors influencing disease outcome during the first year of treatment, especially TS1 versus TS2.
* To determine total, medical and non-medical costs, during the first year of treatment and to compare these costs between patients treated according TS1 versus TS2.

Exploratory objectives

- To sequentially evaluate several blood biomarkers, including anti-BP180 and anti-BP230 IgG autoantibodies, IL-17, IL-23, IL-12 or other biologic makers and to compare them according the treatment scheme (TS1 versus TS2).

Included patients with bullous pemphigoid will be followed for 1 year. Baseline and 6 follow-up visits are planned to record disease activity, treatment and laboratory monitoring modalities and to collect blood samples for ancillary studies. Clinical data recorded at baseline are gender, age and associated medical conditions (neurological disorders: dementia, stroke, Parkinson's disease, multiple sclerosis; malignancy; other diseases). Baseline clinical evaluation includes the number of daily new blisters for 3 consecutive days, localization of skin or mucous membrane blisters and erosions and BPDAI (bullous pemphigoid disease area index). Extensive bullous pemphigoid is defined as the occurrence of at least 10 new daily blisters. The first-line treatment used will be recorded (superpotent topical CS, i.e. clobetasol propionate cream, 20-30g per day; methotrexate; other systemic therapy). At each visit, the presence of pruritus, erythematous or eczematous or urticarial plaques, and the number of new daily blisters are recorded and a BPDAI (bullous pemphigoid disease area index) is calculated. Topical and systemic treatments for bullous pemphigoid are recorded at each visit, as the occurrence and date of relapse, which eventually occurred. Relapse is defined as the reappearance of ≥3 new daily blisters along with pruritus and/or erythematous, eczematous or urticarial plaques.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient or a legally authorized representative person.
* Patients affiliated to social security system
* BP newly diagnosed according to the following criteria: i) suggestive clinical features; ii) histological picture of subepidermal blisters with an infiltrate of eosinophils in the superficial dermis; iii) presence of continuous, linear deposits of IgG and C3 deposits along the skin basement membrane zone by direct IF.
* Patients: no prior superpotent topical steroid therapy or systemic treatment for BP for more than 2 weeks

Exclusion Criteria:

* BP in relapse
* Pemphigoid of pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with bullous pemphigoid
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
BPDAI (bullous pemphigoid disease area index) | up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France